CLINICAL TRIAL: NCT01783067
Title: Zinc and Iron Bioavailability From Bio-fortified Pearl Millet
Brief Title: Zinc and Iron Bioavailability From Biofortified Pearl Millet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Jawaharlal Nehru Medical College (Other); HarvestPlus (Other); International Atomic Energy Agency (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 13-1430
Record Dates: First submitted 2013-01-28; First posted 2013-02-04 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Nutritional Deficiency
Keywords: Biofortification; Pearl millet; Iron absorption; Zinc absorption
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Iron and zinc biofortified pearl millet (Experimental): Participants in the experimental arm consume pearl millet which has been biofortified with iron and zinc.
  Interventions: Other: Biofortified pearl millet
- Pearl millet (Active Comparator): Participants in the control arm consume non-biofortified pearl millet.
  Interventions: Other: Pearl millet

INTERVENTIONS:
Other: Pearl millet — Participants in the control arm consume pearl millet which has not been biofortified. The intervention is consumed for two days.
  Arms: Pearl millet
Other: Biofortified pearl millet — Participants in the experimental arm consume pearl millet biofortified with iron and zinc. The intervention is consumed for two days.
  Arms: Iron and zinc biofortified pearl millet

SUMMARY:
Populations who consume non-fortified plant-based diets are at increased risk of iron and zinc deficiencies. The purpose of this randomized controlled study is to determine the absorption of iron and zinc from pearl millet biofortified with these two micronutrients. Forty children aged 2 years in Kanartaka, India are randomized to consume biofortified pearl millet (Group 1) or control pearl millet (Group 2) for two days. Quantities of zinc and iron absorbed are measured with established stable isotope extrinsic labeling techniques and analyses of duplicate diets.

DETAILED DESCRIPTION:
Nutritional deficiency of iron in 30-70% of young children in different communities in India is well documented and has proved challenging to eradicate both in India and globally. Less is known about zinc deficiency, but zinc and iron are generally present in the same foods and there is also growing evidence for the public health importance of zinc deficiency in young children on a global basis. In populations that depend primarily on plant-based foods, biofortification of major food staples by traditional selective plant breeding procedures offers an attractive strategy for preventing iron and zinc deficiency in all age groups. Pearl millet, a major food staple in several areas of India, has both naturally relatively high concentrations of iron and zinc with demonstrated potential to increase these levels further with plant breeding. Before embarking on complex, costly efficacy, effectiveness studies of the potential health benefits of this biofortified grain, the objective of this project is to determine the extent to which iron and zinc absorption is increased in very young children who consume pearl millet as the primary grain and major food staple. This is a short term, cross-sectional double-blinded study in which the test or control pearl millet is fed for a total of 9 days. Primary outcome measures are the increases in iron and zinc absorption over a two-day period. Test meals will be labeled with a zinc stable isotope on Day 8 and an iron stable isotope on Days 8 and 9 during which days participants and their mothers will stay in their community health center. Food intake will be weighed and duplicate diets obtained. Percentage iron absorption will be determined from erythrocyte enrichment on Day 23. Fractional zinc absorption will be measured from urine enrichment with orally and intravenously administered zinc isotopes from timed samples collected on Days 12-15. Daily absorption of these minerals will be determined. Increases in intake and absorption of these minerals (mg/d) will be evaluated with respect to estimated dietary and physiologic requirements.

ELIGIBILITY:
Inclusion Criteria:

* lives in one of the targeted communities
* apparently healthy
* 23 m of age [may need modification]
* Hemoglobin (Hb) > 8 g/dl
* ferritin ≤ 12mg/L

Exclusion Criteria:

* Hemoglobin (Hb) < 8g/dl
* serum ferritin > 12 (even after correction for C-reactive protein (CRP)/ Alpha Glyco Protein (AGP)
* thalassemia
* birth weight < 2,500 g
* birth defect affecting growth and development
* chronic infection

Ages: 18 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2011-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Absorption of iron from pearl millet | 2 days
  Absorption of iron will be measured while the participants are eating pearl millet as their major food staple which will provide at least 50% energy and at least 75% iron, zinc and phytate of the diet. Fractional absorption of iron for two days will be measured by extrinsic labeling with stable isotopes of iron and measuring erythrocyte enrichment. Measurement of total iron in duplicate diets on test days will allow determination of quantity of this micronutrient absorbed (mg/d).
Absorption of zinc from pearl millet | 1 day
  Absorption of zinc will be measured while the participants are eating pearl millet as their major food staple which will provide at least 50% energy and at least 75% iron, zinc and phytate of the diet. Fractional absorption of zinc for a day will be measured by extrinsic labeling with stable isotopes of zinc. Fractional absorption of zinc will be measured by a dual isotope tracer ratio technique. Measurement of total zinc in duplicate diets on test day will allow determination of quantity of this micronutrient absorbed (mg/d).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hambidge, MD, Principal Investigator — University of Colorado, Denver
Locations (2):
- University of Colorado Denver, Aurora, Colorado, United States
- JN Medical College (Human field studies), Belagavi, Karnataka, India

REFERENCES:
- [Background] Kodkany BS, Bellad RM, Mahantshetti NS, Westcott JE, Krebs NF, Kemp JF, Hambidge KM. Biofortification of pearl millet with iron and zinc in a randomized controlled trial increases absorption of these minerals above physiologic requirements in young children. J Nutr. 2013 Sep;143(9):1489-93. doi: 10.3945/jn.113.176677. Epub 2013 Jul 10. PMID 23843474
- [Background] Miller LV, Hambidge KM, Krebs NF. Zinc Absorption Is Not Related to Dietary Phytate Intake in Infants and Young Children Based on Modeling Combined Data from Multiple Studies. J Nutr. 2015 Aug;145(8):1763-9. doi: 10.3945/jn.115.213074. Epub 2015 Jun 24. PMID 26108545